CLINICAL TRIAL: NCT04643041
Title: Watch and Wait in Patients With dMMR/MSI-H Distal Rectal Cancer Accessed Pathological Complete Response After PD-1 Monoclonal Antibody Therapy-an Open Label, Multicenter, Prospective Study (BASKET)
Brief Title: Watch and Wait in PD-1 Monoclonal Antibody Treated dMMR/MSI-H Distal Rectal Cancer
Acronym: BASKET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2020132
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer
Keywords: PD-1 monoclonal antibody; watch and wait; dMMR/MSI-H; distal rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: patients with DNA mismatch repair-deficient or microsatellite instability-high distal rectal cancer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- watch and wait (Experimental): patients with DNA mismatch repair-deficient or microsatellite instability-high distal rectal cancer accessed pathological complete response after 6 courses of PD-1 monoclonal antibody (200mg/Course/Q3W) therapy and start watch and wait.
  Interventions: Behavioral: watch and wait

INTERVENTIONS:
Behavioral: watch and wait — patients with DNA mismatch repair-deficient or microsatellite instability-high distal rectal cancer accessed pathological complete response after 6 courses of PD-1 monoclonal antibody (200mg/Course/Q3w) therapy and start watch and wait.

SUMMARY:
Immunotherapy has achieved significant therapeutic effect in DNA mismatch repair-deficient or microsatellite instability-high (dMMR/MSI-H) colorectal cancer (CRC) , more than fifty percent of dMMR/MSI-H CRC patients might get pathological complete response(pCR) after PD-1 monoclonal antibody treatment. For distant rectal cancer(RC), radical resection and neoadjuvant chemotherapy or chemoradiotherapy might cause lots of treatment cost,damage to defecation and sexual function, acute toxicity, chronic dysfunction, even loss of anus and psychological disorder. This study aims to evaluate the effect and safety of watch and wait in patients with dMMR/MSI-H distal RC accessed pCR after PD-1 monoclonal antibody therapy.

DETAILED DESCRIPTION:
Immunotherapy has achieved significant therapeutic effect in DNA mismatch repair-deficient or microsatellite instability-high (dMMR/MSI-H) colorectal cancer (CRC). MMR expression and MSS status are the important effective factors of immunotherapy. PD-1monocolnal antibody therapy has accessed excellent treatment effect in advanced dMMR/MSI-H CRC and neoadjuvant therapeutic effect in early colon cancer, more than fifty percent of dMMR/MSI-H CRC patients might get pathological complete response(pCR) after PD-1 monoclonal antibody treatment. The treatments had been proved to be safe and the toxicities were controllable. Rectal cancer(RC) is one of the most common malignant tumors in China. So far, radical resection with or without neoadjuvant chemotherapy of chemoradiotherapy are still standard comprehensive treatments recommended to distal RC by NCCN, ESMO and CSCO. For distant RC, radical resection and neoadjuvant chemotherapy or chemoradiotherapy might cause lots of treatment cost,damage to defecation and sexual function, acute toxicity, chronic dysfunction, even loss of anus and psychological disorder. So far, whether watch and wait could be performed in patients with dMMR/MSI-H distal RC accessed pCR after PD-1 monoclonal antibody therapy or not is still not clear. Thus, this study aims to evaluate the effect and safety of watch and wait in patients with dMMR/MSI-H distal RC accessed pCR after PD-1 monoclonal antibody therapy.

ELIGIBILITY:
Inclusion Criteria:

Preliminary inclusion criteria：

* Histological identified rectal adenocarcinoma,
* Tumor biopsy immunohistochemical (IHC) identified dMMR, including one or more deficient of the MSH1,MSH2,MSH6 and PMS2 protein expression and diagnosed as deficient mismatch repair(dMMR), or next generation sequencing identified (MSI-H)； MRI identified tumor inferior margin lower than peritoneal reflection,
* Clinical staging TxNxM0, with or without positive MRF, with or without positive EMVI,
* Staging method：all patients undergo rectal palpation, high resolution MRI ± transrectal Ultrasound examination，positive perienteric lymph node(LN): short diameter ≥10mm LN or LN with typical metastatic shape and MRI character, clinical data should be re-evaluated and judged by center evaluation group when there are contradictory stagings，distant metastasis were excluded by chest and abdominal enhanced CT and pelvic enhanced MRI,
* No intestinal obstruction symptom，or obstruction relieved after proximal colostomy,
* No rectal surgery history,
* No chemotherapy or radiotherapy history,
* No biopharmaceutical treatment history(such as monoclonal antibody), immunotherapy(such as anti PD-1antibody, anti PD-L1 antibody, anti PD-L2 antibody or anti CTLA-4), or other research drug treatment,
* Endocrinotherapy history restriction:No
* Informed consent assigned, Final inclusion criteria：
* Clinical complete response (cCR)(Chest,abdominal and pelvic enhanced CT or pelvic enhanced MRI or transrectal ultrasound proved)
* Transrectal ultrasound biopsy or endoscopic biopsy proved pathologically complete response (pCR)

Exclusion Criteria:

* Arrhythmia need anti-arrhythmia treatment(except β-blocking agent or Digoxin)，symptomatic coronary heart disease or myocardial ischemia(myocardial infarction within 6 months) or congestive heart-failure (CHF) > NYHA grade II,
* Severe hypertension not well controlled by drugs,
* HIV infection history or active phase of chronic Hepatitis B or C(high copies of virus DNA),
* Active tuberculosis(TB)，accepting anti-TB treatment or anti-TB treatment within 1 year before trial screen,
* Other active clinical severe infection(NCI-CTC V5.0),
* Outside pelvic distant metastasis evidences,
* Dyscrasia, organ dysfunction,
* Pelvic or abdominal radiotherapy history,
* Multiple CRC or Multi-primary tumors；
* Epilepsy need treatments(Steroid or anti-epilepsy therapy),
* Other malignant tumor history within 5 years,
* Over abuse of drugs, medical and psychological or social conditions that might interfere patients or evaluation of the study results,
* Any active autoimmune disease or autoimmune disease history (including but not restricted：interstitial pneumonia, uveitis,enteritis, hepatitis,hypophysitis, nephritis, hyperthyroidism, hypothyroidism, asthma need bronchodilators),
* Any anti-infection vaccine injection 4 weeks before inclusion ,
* Long-term exposure to immune-suppressor, combination of systemic or topical use of corticosteroids (dose>10mg/day prednisolone or equivalent hormone)；
* Known or suspicious allergy to any study related drugs,
* Any unstable state might cause damage to the safety and compliance of patients,
* Pregnant or breast feeding women who has ability to have children while without contraception,
* Refuse to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
1 year DFS rate | 1 year
  1 year Disease Free Survival Rate

SECONDARY OUTCOMES:
Incidence rate of Grade ≥3 PD-1monoclonal antibody-related adverse events | 1 year
  Incidence rate of participants with Grade ≥3 PD-1monoclonal antibody-related adverse events as assessed by CTCAE v4.0
local recurrent rate | 3 years
  local recurrent rate of original rectal cancer
distant metastasis rate | 3 years
  distant metastasis rate
3 years DFS Rate | 3 years
  3 years Disease Free Survival Rate
3 years OS rate | 3 years
  3 years Overall Survival Rate

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Wang, MD, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University; Jun Huang, MD, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sun Yatsen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott E. Chemohormonal therapy in metastatic hormone-sensitive prostate cancer. Sweeney CJ, Chen YH, Carducci M, Liu G, Jarrard DF, Eisenberger M, Wong YN, Hahn N, Kohli M, Cooney MM, Dreicer R, Vogelzang NJ, Picus J, Shevrin D, Hussain M, Garcia JA, DiPaola RS. Department of Medicine; Department of Biostatistics and Computational Biology; Dana-Farber Cancer Institute, Boston; Harvard Medical School, Boston; Johns Hopkins University, Baltimore; University of Wisconsin Carbone Cancer Center; School of Medicine and Public Health; Madison; Fox Chase Cancer Center, Temple University Health System, Philadelphia; Indiana University Melvin and Bren Simon Cancer Center, Indianapolis; Mayo Clinic, Rochester, MN; University Hospitals Case Medical Center, Seidman Cancer Center; Cleveland Clinic Taussig Cancer Institute; Both in Cleveland; University of Virginia Cancer Center, Charlottesville; Comprehensive Cancer Centers of Nevada, Las Vegas; Siteman Cancer Center, Washington University School of Medicine, St. Louis; NorthShore University Health System, Evanston, IL; University of Michigan Comprehensive Cancer Center, Ann Arbor; Rutgers Cancer Institute of New Jersey, New Brunswick.N Engl J Med. 2015 Aug 20;373(8):737-46. [Epub 2015 Aug 5]. doi: 10.1056/NEJMoa1503747. Urol Oncol. 2017 Mar;35(3):123. doi: 10.1016/j.urolonc.2016.12.021. Epub 2017 Feb 1. PMID 28159490
- [Background] Sclafani F. PD-1 inhibition in metastatic dMMR/MSI-H colorectal cancer. Lancet Oncol. 2017 Sep;18(9):1141-1142. doi: 10.1016/S1470-2045(17)30512-0. Epub 2017 Jul 19. No abstract available. PMID 28734760
- [Background] Das R, Verma R, Sznol M, Boddupalli CS, Gettinger SN, Kluger H, Callahan M, Wolchok JD, Halaban R, Dhodapkar MV, Dhodapkar KM. Combination therapy with anti-CTLA-4 and anti-PD-1 leads to distinct immunologic changes in vivo. J Immunol. 2015 Feb 1;194(3):950-9. doi: 10.4049/jimmunol.1401686. Epub 2014 Dec 24. PMID 25539810
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Prasad V, Kaestner V, Mailankody S. Cancer Drugs Approved Based on Biomarkers and Not Tumor Type-FDA Approval of Pembrolizumab for Mismatch Repair-Deficient Solid Cancers. JAMA Oncol. 2018 Feb 1;4(2):157-158. doi: 10.1001/jamaoncol.2017.4182. No abstract available. PMID 29285544